CLINICAL TRIAL: NCT05633927
Title: Prospective Study to Evaluate the Persistence and Characteristics of Humoral and Cellular Immunity Against SARS-COV-2 After Vaccination in HIV-infected Patients Severely Immunosuppressed
Brief Title: Humoral and Cellular Immunity Against SARS-COV-2 Vaccine in HIV-infected Patients Immunosuppressed
Status: Completed | Type: Observational
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Luis F. Lopez-Cortes, Principal Investigator, Hospitales Universitarios Virgen del Rocío
Other Study IDs: CoVa-VIH-2021
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: SARS-CoV-2 RNA Vaccines; HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-immunological responder: Patients who start ART with <350 CD4+ T cells, maintaining undetectable viral load, and increasing <200 CD4+ T cell count after 18 months of follow-up.
  Interventions: Biological: SARS-CoV-2 Vaccine
- Immunological responder: Patients with >350 CD4+ T cells
  Interventions: Biological: SARS-CoV-2 Vaccine

INTERVENTIONS:
Biological: SARS-CoV-2 Vaccine — Analyse humoral and cellular response to SARS-CoV-2 Vaccine.

SUMMARY:
Prospective, non-equality, cohort study, where investigators propose to analyze humoral and cellular immunity after two doses of SARS-CoV-2 RNA vaccines in HIV-infected participants severely immunosuppressed.

A total of 92 HIV-infected subjects over 18 years old with ≤200 CD4/μl (experimental group; n=46) and ≥ 350 CD4/μl (as control group; n=46) who have completed two doses vaccination against SARS-CoV-2 will be included in the study.

Primary Objectives:

* To analyze the percentage of participants with SARS-CoV-2-specific IgG after 1, 6, and 12 months after vaccination in subjects with ≤200 vs ≥350 CD4/μL by electrochemiluminescence immunoassay (Elecsys® Anti-SARS-CoV-2. Roche Diagnostics).
* To analyze the percentage of subjects with specific T and memory B lymphocyte response against SARS-CoV-2 after 1, 6, and 12 months after vaccination with <200 vs ≥350 CD4/μL. Multiparametric flow cytometry in peripheral blood mononuclear cells (PBMCs) will be performed to detect the production of cytokines (IL-2, TNF-α and IFN-γ), cytolytic (perforin and granzyme B) and degranulation (CD107a) molecules from T cells, as well as to identify memory B cells specific to SARS-CoV-2 IgG+.

Secondary Objectives: To analyze in participants with <200 vs ≥350 CD4/μl after 1, 6, and 12 months after vaccination:

* Quantification of specific IgG titers against SARS-CoV-2
* The association of the T response to SARS-CoV-2 with humoral response parameters.
* The association of the T response against SARS-CoV-2 with other parameters of immune activation, inflammation and immunosenescence. The phenotypes of maturation (CD45RA and CD27), activation (HLA-DR and CD38), senescence (CD57+CD28-) and markers of immune exhaustion (TIGIT, LAG-3, TIM-3 and PD-1) in CD4 and CD8 lymphocytes T will be determined by multiparametric flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected subjects over 18 years old and ≤200 CD4/μl who have completed vaccination against SARS-CoV-2.
2. HIV-infected subjects with ≥350 CD4/μl who have completed vaccination against SARS-CoV-2 matched by age and sex as control group.
3. Sign the informed consent.

Exclusion Criteria:

1. Neoplastic or autoimmune disease known.
2. Treatment with steroids, immunomodulators, interferon, chemotherapy or any pathology that may impact immunological parameters after vaccination against SARS-CoV-2.
3. Active infections at the time of sampling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was designed as a cohort study comparing the immune response after vaccination of HIV-infected subjects with the hypothesis that subjects with ≤200 CD4/μL will have a worse response than those with CD4 count ≥ 350/μL.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Antibodies | 24 months
  Analyse the percentage of subjects with SARS-CoV-2-specific IgG after 1, 6, and 12 months after complete vaccination regimen in HIV-infected subjects and ≤200 vs ≥350 CD4/μL. And to analyse the percentage of subjects with specific T and memory B lymphocyte response against SARS-CoV-2

CONTACTS AND LOCATIONS:
Locations (1):
- Virgen del Rocio University Hospital, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lopez-Cortes LF, Saborido-Alconchel A, Trujillo-Rodriguez M, Serna-Gallego A, Llaves-Flores S, Munoz-Muela E, Perez-Santos MJ, Lozano C, Mejias-Trueba M, Roca C, Espinosa N, Gutierrez-Valencia A. Humoral and cellular immunity to SARS-COV-2 after vaccination with mRNA vaccines in PLWH with discordant immune response. Influence of the vaccine administered. Front Immunol. 2023 Mar 15;14:1129753. doi: 10.3389/fimmu.2023.1129753. eCollection 2023. PMID 37006309
- See also: Related Info — https://www.frontiersin.org/articles/10.3389/fimmu.2023.1129753/full
- See also: Related Info — http://www.frontiersin.org/articles/10.3389/fimmu.2023.1129753/full